CLINICAL TRIAL: NCT02168725
Title: A Phase I, Dose-escalation Study of the Safety, Pharmacokinetics and Efficacy of Weekly Intravenous Briciclib in Patients With Advanced Solid Tumors
Brief Title: Dose-escalation, Safety and Pharmacokinetic Study of Briciclib in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was placed on hold by the FDA due to manufacturing issues and was not restarted.
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 08-02; COMIRB 14-0565 (Other: Univ. of Colorado Denver Multiple Institutional Review Board)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Neoplasms; Advanced Solid Tumor
Keywords: briciclib; Dose escalation; Maximum tolerated dose
MeSH Terms: conditions — Neoplasms | interventions — ON 013105

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- briciclib (Experimental): The starting dose of briciclib in the Escalation Stage will be 17 mg/week, with subsequent dose escalation levels of 35 mg, 70 mg, 140 mg, 280 mg, 560 mg, and 1120 mg. The dose of briciclib in the RPTD Confirmation Stage will be the dose as determined during the escalation stage. At each dose level, briciclib will be administered as a 2-hour intravenous infusion, once-a-week per 3-week cycles.
  Interventions: Drug: briciclib

INTERVENTIONS:
Drug: briciclib
  Other Names: ON 013105

SUMMARY:
The main objectives of this study are to determine the safety profile of briciclib, an experimental anti-cancer drug, as it is administered intravenously once weekly as escalating doses in adult patients with advanced cancer and solid tumors, and to determine the highest dose of briciclib that can be safely given. Secondary objectives are to determine how the amount of briciclib in circulation changes over time and how much briciclib gets into the urine for excretion, and to document potential anti-tumor effects of briciclib.

DETAILED DESCRIPTION:
This will be a Phase I, 2-stage, open-label, dose-escalating, multicenter study of the 2-hour, once-a-week intravenous (IV) administration of briciclib in 3-week cycles, in up to 54 adult patients with advanced cancer and solid tumors. The study will be conducted in 2 stages: a dose-escalation stage to determine the Maximum Tolerated Dose (MTD) and a Recommended Phase 2 Dose (RPTD) confirmation stage. Patients with stable disease (SD) or response may remain treated on study until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed solid tumor (leukemia and lymphoma are excluded)
2. Malignancy that is incurable and for which standard (FDA approved or established standard clinical practice) curative, or palliative measures do not exist or are no longer effective
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
4. Minimum expected life expectancy > 6 months
5. One or more measurable lesion(s) ("target lesion[s]") that can be accurately measured in at least 1 dimension
6. Willing to adhere to the prohibitions and restrictions specified in the protocol
7. The patient must sign an informed consent form (ICF)

Exclusion Criteria:

1. Recent major surgery (within the past 14 days)
2. Chemotherapy or dose of other potentially myelosuppressive treatment within 3 weeks prior to Screening (6 weeks for nitrosoureas or mitomycin C)
3. No more than a total cumulative dose of 450 mg/m^2 of prior doxorubicin chemotherapy
4. Definitive radiotherapy (> 10 fractions and maximal area of hematopoietic active Bone Marrow treated greater than 25%) within 4 weeks prior to Screening
5. Palliative radiotherapy (≤ 10 fractions) within 2 weeks prior to Screening
6. Known brain metastases, except brain metastases that have been previously removed or irradiated and currently have no clinical impact
7. Residual adverse events due to previously administered agents (except alopecia, stable residual neuropathy, and residual hand, foot syndrome) that have not recovered to Grade 1 or below in severity level (based on NCI CTCAE) before Screening
8. Ascites requiring active medical management, including paracentesis
9. Pleural effusion requiring active medical management
10. Peripheral bilateral edema requiring active medical management
11. Hyponatremia (serum sodium value less than 130 mEq/L)
12. History of allergic reactions attributed to compounds of similar chemical or biologic composition to briciclib
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, bleeding, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
14. History of myocardial infarction
15. Any other concurrent investigational agent or chemotherapy, radiotherapy, hormonotherapy, or immunotherapy. Exceptions are long-term hormonals for prostate (eg, goserelin) and octreotide for neuroendocrine malignancies
16. Patients who are positive for human immunodeficiency virus type 1 (HIV-1) and are receiving combination anti-retroviral therapy
17. Hemoglobin (Hgb) < 9 g/dL
18. White Blood Cell count (WBC) < 4,000/µL
19. Absolute Neutrophil Count (ANC) < 1,500/µL
20. Platelet (PLT) count ≤ 100,000/µL
21. Total bilirubin greater than 1.5 x the institutional upper limit of normal (ULN)
22. Aspartate transaminase (AST) or alanine transaminase (ALT) ≥ 2.5 x institutional ULN. If liver function abnormalities are due to metastatic disease, patients are eligible provided the ALT and AST are < 5 x ULN
23. Serum creatinine > 2 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to 1 year
  Adverse events will be grouped by system organ class (SOC) and preferred term (PT) using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA), and will be summarized by worst grade according to NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
Number of patients with Dose Limiting Toxicity (DLT) | Up to 3 weeks
  Dose-limiting toxicity is defined as an adverse event that is considered to be drug-related and meets one of the Protocol definitions.
Maximum Tolerated Dose | 3 weeks
  Maximum Tolerated Dose (MTD) will be defined during the Dose Escalation Stage based on evaluation of the number of patients with Dose-limiting Toxicity (DLT). The MTD will be used to determine the Recommended Phase 2 Dose (RPTD).

SECONDARY OUTCOMES:
Concentration of briciclib in the plasma | 24 hours
  The amount of briciclib in the plasma of patients in the Recommended Phase 2 Dose (RPTD) Confirmation stage only will be measured by a validated Liquid Chromatography-Mass Spectroscopy (LC-MS) method. Pharmacokinetic parameters will be derived from the concentration versus time values.
Concentration of briciclib in the urine | 24 hours
  The amount of briciclib in the urine of patients in the Recommended Phase 2 Dose (RPTD) Confirmation stage only will be measured by a validated Liquid Chromatography-Mass Spectroscopy (LC-MS) method. Pharmacokinetic parameters will be derived from the concentration versus time values.
Change in size of tumors | Up to 1 year
  Change in the overall tumor will be determined from the tumor burden at Baseline following Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

OTHER OUTCOMES:
Biomarker Concentration or Activity | Up to 1 year
  An exploratory objective of this study is to evaluate the biological effect of briciclib on cell-cycle pathways, cyclin D1, and other potential surrogate biomarker(s) of efficacy and/or toxicity in tumor tissue and peripheral blood mononuclear cells (PBMNC).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Jimeno, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Hospital Anschutz Medical Campus, Aurora, Colorado
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee